CLINICAL TRIAL: NCT05559684
Title: Analgesic Efficacy of Bilateral Ultrasound Guided Transversus Thoracic Muscle Plane Block Versus Erector Spinae Plane Block in Pediatric Patients Undergoing Corrective Cardiac Surgeries - A Randomized Controlled Trial
Brief Title: Analgesic Efficacy of Bilateral US Guided TTPB vs ESPB in Pediatric Patients Undergoing Corrective Cardiac Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Engy I. Abueldahab, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: md-61-2022
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Pain, Postoperative
Keywords: Transversus thoracic muscle plane block; Erector spinea plane block; Pediatric cardiac surgery; Multimodal anelgesia in pediatric cardiac surgeries; TTPB; ESPB
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Randomization will be achieved by using an online random number generator. Patient codes will be placed into sequentially numbered sealed opaque envelopes by a research assistant who is not involved in the study. A medical doctor not involved in patient management will be responsible for opening the envelope and give the instructions contained within each envelope to the anesthesiologist who is expert in doing the ESPB in patients included within the block group. This expert anaesthesiologist will not be involved in collecting data but another anaesthesist blinded to the type of block will be responsible for patient management and collecting the intra-operative and postoperative data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): Patients in this group will receive fentanyl infusion at a dose of (0.5 μg/kg/h) all through the whole operation; in addition to
  1μg/kg during skin incision, sternotomy, aortic cannulation and increase in MBP or HR more than 20% of the baseline readings.
- Erector Spinae Plane Block (Active Comparator): This group will receive fentanyl infusion at a dose of (0.5 μg/kg / h) all through the whole operation plus Ultrasound guided bilateral ESPB which will be done by injecting 0.4 ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%) at each side
  Interventions: Procedure: Erector spinae plane block
- Transversus Thoracis Plane Block (Experimental): This group will receive fentanyl infusion at a dose of (0.5 μg/kg / h) all through the whole operation plus ultrasound guided bilateral TTPB which will be done by injecting 0.4 ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%) at each side
  Interventions: Procedure: Transversus thoracis plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — Under strict aseptic precautions, The T3 spinous process will be located. A high-frequency 12 MHz linear US transducer will be placed in a longitudinal orientation 3 cm lateral to the T3 spinous process corresponding to the T2 transverse process. Three muscles; trapezius (uppermost), rhomboids major (middle), and erector spinae (lowermost) will be identified superior to the hyperechoic transverse process. Using in-plane approach a 25 G needle will be inserted in caudal-cephalad direction, until the tip is deep to erector spinae muscle. Correct needle tip location will be confirmed by injecting 3 mL of normal saline and visualizing the linear LA spread (i.e., hydrodissection) in the fascial plane between the erector spinae muscle and the transverse process. Then, 0.4 ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%) will be injected and visualizing the linear LA spread in the fascial plane between the erector spinae muscle and the transverse process.
  Arms: Erector Spinae Plane Block
Procedure: Transversus thoracis plane block — Under strict aseptic precautions, the T4-T5 intercostal space is identified under US using the US probe in the longitudinal plane 1 cm lateral to the sternal border. A high-frequency linear transducer is used. Next, a parasternal sagittal view of the intercostal muscle and the transverses thoracis muscle between the 4th and 5th rib is visualized above the pleura and a 22G, 5-10 cm needle is inserted in-plane (according to patient's body habitus and relevant anatomy) to the transducer with bevel up until the tip of the needle is located in the transverses thoracis muscles. After excluding intravascular and intrapleural placement, local anesthetic is adminstred bilaterally by injecting 0.4ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%) at each side.
  Arms: Transversus Thoracis Plane Block

SUMMARY:
Corrective cardiac surgeries include a bundle of major surgeries that take place in pediatric patients and require imperative perioperative pain control; hence, the art of healing starts from trying to diminish or abolish pain.

The use of highly potent opioids for paediatric cardiac anaesthesia has gained widespread popularity during the last 20 years . In addition to the important advantage of hemodynamic stability, the large-dose opioid-based anaesthetic techniques also blunt the stress response; however, large doses can cause over sedation, respiratory depression and prolonged mechanical ventilation after surgery .

There are many ways to limit pain in such population with the topper potent opioids in the last several years. But new regional pain management modalities started to arise because of their known effect to diminish neuroendocrine stress response, provide excellent postoperative analgesia, and facilitate early postoperative extubation .

Of the new evolving methods, the bilateral Transversus Thoracic Muscle Plane Block (TTPB) provides analgesia to the anterior chest wall and proved to be efficient in pediatric patients undergoing cardiac surgery using a median sternotomy approach .

The bilateral Erector Spinae Plane Block (ESPB) is also one of the recently known pain controlling techniques used in pediatric cardiac surgeries. It became popular because it is much safer and easily administered than other alternative regional techniques as thoracic paravertebral and thoracic epidural block .

DETAILED DESCRIPTION:
I. Study design and randomization

Our study will be designed to estimate the analgesic effect of single shot bilatral transversus thoracic muscle plane block compared to that of erector spinae plane block in pediatric patients undergoing corrective cardiac surgeries including atrial septal defect (ASD) repair, ventricular septal defect (VSD) repair, atrioventricular (AV) canal repair, Glenn procedure, Fontan procedure and subaortic membrane resection. Our primary outcome will be the total dose of intra-operative fentanyl boluses.

Randomization will be achieved by using an online random number generator. Patient codes will be placed into sequentially numbered sealed opaque envelopes by a research assistant who is not involved in the study. A medical doctor not involved in patient management will be responsible for opening the envelope and give the instructions contained within each envelope to the anesthesiologist who is expert in doing the ESPB in patients included within the block group. This expert anaesthesiologist will not be involved in collecting data but another anaesthesist blinded to the type of block will be responsible for patient management and collecting the intra-operative and postoperative data.

II. Study setting and location

The study will be conducted in the pediatric cardiothoracic operation theatre in Abu El Reesh Pediatric Hospital - Cairo University.

III. Study population

The study will be conducted on pediatric patients aged 2 months - 4 years, ASA II and III undergoing corrective cardiac surgeries (with midline sternotomy incision). The patients will be randomly assigned to one of 3 groups Group (A): (Control group): This group will receive fentanyl infusion at a dose of (0.5 μg/kg/h) all through the whole operation .

Group (B): This group will receive fentanyl infusion at a dose of (0.5 μg/kg/h) all through the whole operation plus Ultrasound guided bilateral ESPB which will be done by injecting 0.4 ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%) at each side .

Group (C): This group will receive fentanyl infusion at a dose of (0.5 μg/kg/h) all through the whole operation plus ultrasound guided bilateral TTPB which will be done by injecting 0.4 ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%) at each side .

IV. Study Procedures

-Preoperative:-

All patients will attend at the pre- anesthesia room with their parents 1 hour before the procedure after taking approval of research ethical committee and informed consent.

Detailed history from the parents will be taken followed by a full and detailed clinical examination of the child then all investigations including CBC, coagulation profile, liver enzymes, kidney function tests, CXR, echocardiography/cardiac catheterization and blood grouping will be checked.

-Intraoperative:-

Non-invasive blood pressure, pulse oximetry and ECG will be applied to all patients. All patients will be premedicated by intramuscular midazolam 2mg/Kg and atropine 0.2 mg/Kg 20 minutes before induction of anesthesia.

Anesthesia will be induced in all patients by sevoflurane5% in 50% O2 followed by placement of peripheral I.V cannula and IV administration of fentanyl (0.5 µg/kg). Oral endotracheal intubation will be facilitated by IV atracurium 0.5 mg/kg and then capnogram will be connected to monitor End-tidal CO2 and muscle relaxation will be maintained by atracurium infusion in a dose of 0.5 mg/ kg/ hr.

All patients will be mechanically ventilated using pressure controlled mode with FiO2 50%, PEEP 5 cmH2O, I : E ratio of 1:2, peak inspiratory pressure (PIP) will be set to deliver a tidal volume of 6-8 ml/kg and respiratory rate will be 15 to 35 cycle / minute according to the age. Our aim is to keep end tidal CO2 between 30-40 mmHg. Isoflurane will be used for maintenance of anaesthesia.

After insertion of a central venous catheter and an arterial cannula, nasopharyngeal temperature probe will be placed.

Patients in Group A will receive fentanyl infusion at a dose of (0.5 μg/kg/h) all through the whole operation.

Patients in Group B will receive fentanyl infusion at a dose of (0.5 μg/kg/h) in addition to ultrasound guided bilateral erector spinae plane block by injecting 0.4ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%) at each side as follows :

Under strict aseptic precautions, The T3 spinous process will be located by palpating and counting down from the C7 spinous process.

A high-frequency 12 MHz linear ultrasound transducer will be placed in a longitudinal orientation 3 cm lateral to the T3 spinous process corresponding to the T2 transverse process.

Three muscles; trapezius (uppermost), rhomboids major (middle), and erector spinae (lowermost) will be identified superior to the hyperechoic transverse process.

Using in-plane approach a 25 G needle will be inserted in caudal-cephalad direction, until the tip is deep to erector spinae muscle.

Correct needle tip location will be confirmed by injecting 3 mL of normal saline and visualizing the linear LA spread (i.e., hydrodissection) in the fascial plane between the erector spinae muscle and the transverse process.

Now, 0.4 ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%) will be injected and visualizing the linear LA spread (i.e., hydrodissection) in the fascial plane between the erector spinae muscle andthe transverse process.

Patients in Group C will receive fentanyl infusion at a dose of (0.5 μg/kg/h) plus ultrasound guided bilateral transversus thoracic muscle plane block by injecting 0.4ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%) at each side as follows :

Under strict aseptic precautions, the T4-T5 intercostal space is identified under US using the US probe in the longitudinal plane 1 cm lateral to the sternal border. A high-frequency linear transducer is used.

Next, a parasternal sagittal view of the intercostal muscle and the transverses thoracis muscle between the 4th and 5th rib is visualized above the pleura and a 22G, 5-10 cm needle is inserted in-plane (according to patient's body habitus and relevant anatomy) to the transducer with bevel up until the tip of the needle is located in the transverses thoracis muscles.

After excluding intravascular and intrapleural placement, local anesthetic is adminstred bilaterally by injecting 0.4ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%) at each side.

After 15 min, skin incision will be started and rescue analgesia by a bolus of (Fentanyl 1mcg/kg) will be given to the patients in each group. If either mean blood pressure (MBP) or heart rate (HR) increased more than 20% of the baseline readings (as recorded 5 minutes after intubation) provided that there is no other cause of these hemodynamic changes such as inadequate anesthesia and surgical complications.

The block will be considered a failed block if the patient will require more than two boluses of fentanyl during the first 30 minutes of the skin incision and this case will be excluded from the study.

-Postoperative:- All patients will be discharged to the pediatric ICU where they will receive paracetamol in a dose of 15 mg/ kg I.V. every 6 hours as a standard protocol in our unit.

Measurement tools:

Intra-operative:

* The total dose of fentanyl will be calculated.
* Vital signs including HR and MBP will be recorded at the following intervals; (T1: baseline reading 5 min after intubation, T2: after skin incision, T3: after sternotomy, T4: after aortic cannulation, T5: after weaning from bypass and T6: after skin closure).

In the Pediatric ICU:

* Time (in minutes) to 1st rescue analgesia post operatively (Fentanyl) which will be defined to be the elapsed time between giving the block and a patient FLACC score (Table 1) equal or more than 4.
* Total consumption of Fentanyl during the 1st 12 hours post operatively will be calculated.
* Haemodynamics including HR and MBP immediately after admission to ICU then at 60 min, 2 hours, 4hours, 8 hours and 12 hours
* The incidence of complications like postoperative vomiting, hematoma formation, itching, local anesthetic toxicity.
* Pain score assessment immediately after admission to ICU then at 60 min, 2 hours, 4hours, 8hours and 12 hours postoperatively by FLACC score

  * How to assess pain using FLACC score:

    1. Face

       ● Score 0 point if patient has a relaxed face, eye contact and interest in surroundings
       * Score 1 point if patient has a worried look to face, with eyebrows lowered, eyes partially closed, cheeks raised, mouth pursed
       * Score 2 points if patient has deep furrows in the forehead, with closed eyes, open mouth and deep lines around nose/lips
    2. Legs

       ● Score 0 points if patient has usual tone and motion to limbs (legs and arms)
       * Score 1 point if patient has increase tone, rigidity, tense, intermittent flexion/extension of limbs
       * Score 2 points if patient has hyper tonicity, legs pulled tight, exaggerated flexion/extension of limbs, tremors.
    3. Activity

       ● Score 0 points if patient moves easily and freely, normal activity/restrictions

       ● Score 1 point if patient shifts positions, hesitant to move, guarding, tense torso, pressure on body part

       ● Score 2 points if patient is in fixed position, rocking, side-to-side head movement, rubbing body part.
    4. Cry

       ● Score 0 points if patient has no cry/moan awake or asleep

       ● Score 1 point if patient has occasional moans, cries, whimpers, sighs

       ● Score 2 points if patient has frequent/continuous moans, cries, grunts.
    5. Consolability ● Score 0 points if patient is calm and does not require consoling ● Score 1 point if patient responds to comfort by touch or talk in ½- 1 minute

       * Score 2 points if patient requires constant comforting or unable to console. Pain was assessed by the pediatric observational 10-point scale "Face, Leg, Activity, Cry, Consolability (FLACC) pain score.and if the patient FLACC score equal or more than 4, he will receive morphine i.v 0.1mg /kg .

ELIGIBILITY:
Inclusion Criteria:

* Age: 2 months - 4 years.
* ASA II and III.
* Patients undergoing corrective cardiac surgeries with midline sternotomy incision.

Exclusion Criteria:

* Patients whose parents or legal guardians refusing to participate.
* Preoperative mechanical ventilation.
* Preoperative inotropic drug infusion.
* Known or suspected coagulopathy.
* Known or suspected allergy to any of the studied drugs.
* Severe pulmonary hypertension.
* Cardiopulmonary bypass time more than 90 minutes.
* Aortic cross-clamp time more than 45 minutes.
* Total time from induction till ICU transfer more than 4 hours and 30 mins.

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
The total dose of intraoperative fentanyl | All through the surgery
  Amount of fentanyl required by patients in each group

SECONDARY OUTCOMES:
Pain assessment | Immediately after admission to ICU then at 60 min, 2 hours, 4 hours, 8 hours and 12 hours postoperatively
  FLACC score
Intra and postoperative haemodynamics including HR and MBP | Intraoperative T1: baseline reading 5 min after intubation, T2: after skin incision, T3: after sternotomy, T4: after aortic cannulation, T5: after weaning from bypass and T6: after skin closure then Immediately after admission to ICU, 1,2,4,8,12 hours
  Measurement of HR and MBP
Total consumption of Fentanyl during the 1st 12 hours post operatively | Immediately after admission to ICU then at 60 min, 2 hours, 4 hours, 8 hours and 12 hours postoperatively
  Total dose of Fentanyl
Time (in minutes) to 1st rescue analgesia (Fentanyl) post operatively | First 12 hours postoperatively
  The elapsed time between giving the block and a patient FLACC score equal or more than 4
Time of extubation | First 12 hours postoperatively
  Time needed for the patient's condition to be ready for extubation
The incidence of complications | First 12 hours postoperatively
  postoperative vomiting, hematoma formation, itching, local anesthetic toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Amel H Abo Elela, Professor, Study Chair — Cairo University; Mohamed F Youssef, Professor, Study Director — Cairo University; Mai A Madkour, Professor, Study Director — Cairo University; Ahmed A Gado, Lecturer, Study Director — Cairo University
Locations (1):
- Abu Elrish hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
IPD collected in this study, including data dictionaries will be released to other researchers after the end of the study.
  All collected IPD, Study Protocol, Statistical Analysis Plan, Informed Consent Form, Clinical Study Report, Analytic Code all IPD that underlie results in a publication will be available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: November 2022 - November 2023
Access Criteria: URL

REFERENCES:
- [Derived] Madkour MAFA, Abueldahab EIB, Elela AHA, Youssef MF, Gado AA. Analgesic Efficacy of Bilateral Ultrasound-Guided Transversus Thoracic Muscle Plane Block Versus Erector Spinae Plane Block in Pediatric Patients Undergoing Corrective Cardiac Surgeries: A Randomized Controlled Study. J Cardiothorac Vasc Anesth. 2025 Jun;39(6):1495-1505. doi: 10.1053/j.jvca.2025.03.001. Epub 2025 Mar 3. PMID 40122711